CLINICAL TRIAL: NCT00116688
Title: An Open Label Study Evaluating the Safety and Efficacy of Long-Term Dosing of AMG 531 in Thrombocytopenic Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Brief Title: Open Label Extension Study of Romiplostim (AMG 531) in Thrombocytopenic Patients With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030213
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2011-04-06 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-11

CONDITIONS: Thrombocytopenia; Idiopathic Thrombocytopenic Purpura
Keywords: Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenic
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic | interventions — romiplostim

ARMS (1):
- Romiplostim (Experimental): Romiplostim weekly subcutaneous dosing based on screening weight and platelet count. Starting dose of 1 µg/kg up to a maximum dose of 10 µg/kg.
  Interventions: Biological: Romiplostim

INTERVENTIONS:
Biological: Romiplostim — Romiplostim is supplied in a 5 mL single use glass vial as a sterile, white, preservative-free, lyophilized powder.
  Other Names: AMG 531; Nplate

SUMMARY:
The purpose of this study is to determine the safety of romiplostim as a long-term treatment in thrombocytopenic subjects with ITP, to evaluate the long-term platelet response to romiplostim, and to evaluate changes in patient reported outcomes due to the use of romiplostim. Participants must have previously completed a romiplostim ITP study.

ELIGIBILITY:
Inclusion Criteria:

* Must have previously completed a romiplostim ITP study
* Platelet count ≤ 50 x 10 ^9/L
* Written informed consent

Exclusion Criteria:

* Bone marrow stem cell disorder or new active malignancies diagnosed since enrollment in the previous romiplostim ITP study
* Received any alkylating agents within 4 weeks before screening visit or anticipated use during the time of the proposed study
* Currently enrolled in or has not yet completed at least 4 weeks since ending device or drug trial(s) (other than the previous romiplostim ITP study), or subject is receiving other investigational agent(s) other than romiplostim
* Not using adequate contraceptive precautions
* Not available for follow-up assessments
* Has any kind of disorder that compromises the ability of the participant to give informed consent and does not have a legally-acceptable representative and/or is unable to comply with study procedures.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2004-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bussel JB, Kuter DJ, Pullarkat V, Lyons RM, Guo M, Nichol JL. Safety and efficacy of long-term treatment with romiplostim in thrombocytopenic patients with chronic ITP. Blood. 2009 Mar 5;113(10):2161-71. doi: 10.1182/blood-2008-04-150078. Epub 2008 Nov 3. PMID 18981291
- [Background] Kuter DJ, Bussel JB, Newland A, Baker RI, Lyons RM, Wasser J, Viallard JF, Macik G, Rummel M, Nie K, Jun S. Long-term treatment with romiplostim in patients with chronic immune thrombocytopenia: safety and efficacy. Br J Haematol. 2013 May;161(3):411-23. doi: 10.1111/bjh.12260. Epub 2013 Feb 22. PMID 23432528
- [Background] Terrell D, George J, Bussel J, Lyons R, Pullarkat V, Redner R, Nie, Selleslag D, Nie K, Woodard P.Home administration of romiplostim by patients with chronic immune thrombocytopenia (ITP).Journal-001500;
- [Background] Terrell D, George J, Bussel J, Lyons R, Pullarkat V, Redner R, Nie, Selleslag D, Nie K, Woodard P.Home administration of romiplostim by patients with chronic immune thrombocytopenia (ITP).Journal-001752;
- [Derived] Kuter DJ, Mufti GJ, Bain BJ, Hasserjian RP, Davis W, Rutstein M. Evaluation of bone marrow reticulin formation in chronic immune thrombocytopenia patients treated with romiplostim. Blood. 2009 Oct 29;114(18):3748-56. doi: 10.1182/blood-2009-05-224766. Epub 2009 Aug 11. PMID 19671919
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 2 August 2004 through 15 April 2009
Groups:
- Romiplostim in Adults: Romiplostim administered to adult participants subcutaneously weekly at doses up to 30 µg/kg based on platelet counts. After Amendment 1 the maximum weekly dose was reduced to 15 µg/kg, and after Amendment 2 the maximum weekly dose was reduced to 10 µg/kg. However, participants enrolled prior to Amendment 2 who were receiving >10 µg/kg were permitted to remain on that higher dose, but could not increase their dose. In addition, if the participant's dose was decreased, it could not be increased to >10 µg/kg.
- Romiplostim in Pediatric Population: Romiplostim administered to pediatric participants subcutaneously weekly at doses up to 10 µg/kg based on platelet counts.
Period: Overall Study
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population
Started | 292 | 21
Received Study Medication | 291 | 20
Completed | 200 | 17
Not Completed | 92 | 4
Not completed — Protocol deviation | 1 | 0
Not completed — Noncompliance | 3 | 1
Not completed — Adverse Event | 11 | 0
Not completed — Withdrawal by Subject | 26 | 2
Not completed — Requirement for alternative therapy | 11 | 1
Not completed — Physician Decision | 7 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 15 | 0
Not completed — Protocol-specified criteria | 3 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Other | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population | Total
Number analyzed (Participants) | 292 | 21 | 313
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (16.9) | 10.2 (5.1) | 51.3 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 6 | 190
  Male | 108 | 15 | 123
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 13 | 3 | 16
  White or Caucasian | 246 | 13 | 259
  Hispanic or Latino | 21 | 4 | 25
  Asian | 9 | 0 | 9
  Japanese | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Participants with one or more occurrences of one or more adverse events up to 8 weeks after the end of treatment. Participants with more than one event were only counted once.
Time Frame: Duration of treatment plus 8 weeks (up to 285 weeks)
Population: Safety Analysis Set, composed of all participants who received at least one dose of romiplostim
Measure: Number; unit: Participants
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population
Number analyzed (Participants) | 291 | 20
Participants | 284 | 19

2. Secondary Outcome: Number of Participants With a Platelet Response
Description: Platelet response was defined as having a platelet count of ≥ 50 x 10^9/L at any time on study, excluding platelet counts within 8 weeks after receiving any rescue medications.
Time Frame: Duration of treatment (up to 277 weeks)
Population: Efficacy Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Number; unit: Participants
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population
Number analyzed (Participants) | 291 | 20
Participants | 275 | 20

3. Secondary Outcome: Number of Participants With a Reduction or Discontinuation of Concurrent ITP Therapies
Description: The number of participants with a reduction or discontinuation of concurrent immune (idiopathic) thrombocytopenic purpura (ITP) therapies (corticosteroids, danazol, azathioprine) during the study.
Time Frame: Duration of treatment (up to 277 weeks)
Population: Subset of Efficacy Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim and with baseline concurrent ITP therapy.
Measure: Number; unit: Participants
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population
Number analyzed (Participants) | 37 | 2
Participants | 30 | 1

4. Secondary Outcome: Change From Baseline in ITP Patient Assessment Questionnaire
Description: The ITP Patient Assessment Questionnaire (ITP-PAQ) assesses ITP-specific health-related quality of life (HRQOL). This questionnaire assesses ITP specific health-related quality of life (HRQOL). The questionnaire consists of 44 items and has six domains: These domains assess the impact of ITP on Physical Health, Mental Health, Work, Social Activity, Women's Health and Overall QOL. The impact of ITP on Physical Health consists of four sub-scales, which evaluate ITP related Symptoms, Fatigue, Bother and Activity. The impact of ITP on Mental Health consists of two sub-scales, which evaluate Psychological distress and Fear in a population with ITP. Items are scored from 0-100 with higher scores indicating better HRQOL.
Time Frame: Baseline to Week 48
Population: Full analysis set with available data. Patient reported outcomes were only analyzed in adult participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Romiplostim in Adults
Number analyzed (Participants) | 292
scores on a scale
  Physical Health Symptoms (N=209) | 4.20 (13.15)
  Physical Health Fatigue (N=208) | 3.99 (16.00)
  Physical Health Bother (N=204) | 6.43 (17.39)
  Physical Health Activity (N=208) | 5.23 (21.08)
  Emotional Health Psychological (N=208) | 4.01 (15.81)
  Emotional Health Fear (N=209) | 3.48 (12.59)
  Overall Quality of Life (N=210) | 8.32 (19.65)
  Social Quality of Life (N=209) | 3.89 (13.41)
  Women's Reproductive Health (N=71) | 4.51 (16.35)
  Work Quality of Life (N=75) | 2.78 (14.54)

5. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36)
Description: The SF-36 is a widely used generic health-related quality of life measure. It has 36 questions with 8 domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health. Items are scored from 0 to 100 with higher scores indicating better health status.
Time Frame: Baseline to Week 48
Population: Full analysis set with available data. Patient reported outcomes were only analyzed in adult participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Romiplostim in Adults
Number analyzed (Participants) | 292
scores on a scale
  Physical Functioning (N=206) | 1.38 (6.34)
  Role-Physical (N=208) | 2.03 (8.89)
  Bodily Pain (N=206) | 0.94 (7.99)
  General Health Perception (N=208) | 1.31 (7.03)
  Vitality (N=208) | 1.68 (7.47)
  Social Functioning (N=208) | 0.52 (8.21)
  Role-Emotional (N=205) | 1.75 (12.22)
  Mental Health Index (N=208) | 0.91 (7.45)
  Physical Component Summary (N=200) | 1.49 (6.51)
  Mental Component Summary (N=200) | 1.06 (8.80)

6. Secondary Outcome: Change From Baseline in Euroqol-5D (EQ-5D) Index Score
Description: The EQ-5D is a patient-completed, multidimensional measure of health related quality of life. The instrument is applicable to a wide range of health conditions and treatments and results in a single index score and a visual analog scale (VAS) score. The EQ-5D descriptive health profile comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension comprises three levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D health state is defined by combining one level from each of the five dimensions. EQ-5D index values range from -0.59 to 1.00. Higher EQ-5D Index scores represent better health status.
Time Frame: Baseline to Week 48
Population: Full analysis set with available data. Patient reported outcomes were only analyzed in adult participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Romiplostim in Adults
Number analyzed (Participants) | 154
scores on a scale | 0.03 (0.16)

7. Secondary Outcome: Change From Baseline in Euroqol-5D (EQ-5D) Visual Analogue Scale (VAS)
Description: The EQ-5D is a patient-completed, multidimensional measure of health related quality of life. The EQ-5D VAS records the respondent's self-rated health status on a vertical graduated (0-100) visual analogue scale. Higher EQ-5D VAS scores represent better health status.
Time Frame: Baseline to Week 48
Population: Full analysis set with available data. Patient reported outcomes were only analyzed in adult participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Romiplostim in Adults
Number analyzed (Participants) | 150
scores on a scale | 6.05 (14.85)

8. Secondary Outcome: Patient Global Assessment
Description: The Patient Global Assessment is two questions which assess the overall health-related quality of life (HRQOL) and symptoms of the patient. Each item is answered on a 15-point Likert scale ranging from 'A very great deal worse' (1) to 'A very great deal better' (15). A higher score indicates that quality of life or symptoms have improved.
Time Frame: Week 1 and Week 48
Population: Full analysis set with available data. Patient reported outcomes were only analyzed in adult participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Romiplostim in Adults
Number analyzed (Participants) | 292
scores on a scale
  Week 1 (N=271) | 7.61 (2.02)
  Week 48 (N=216) | 8.18 (1.78)

ADVERSE EVENTS:
Time Frame: For adult participants the average duration was 110 weeks; for pediatric participants the average duration is 82 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. One adult patient and one pediatric patient did not receive the investigational product and were not included in the adverse event table.
Arm/Group | Romiplostim in Adults | Romiplostim in Pediatric Population
Serious Adverse Events (participants affected / at risk) | 117/291 | 2/20
Other Adverse Events (participants affected / at risk) | 270/291 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim in Adults (N=291) | Romiplostim in Pediatric Population (N=20)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow disorder (Blood and lymphatic system disorders) | 4 | 0
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 1 | 0
Evans syndrome (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 7 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 4 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 5 | 0
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 2 | 0
Hernia pain (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Mechanical complication of implant (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Candidiasis (Infections and infestations) | 1 | 0
Catheter bacteraemia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Meningitis listeria (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Megakaryocytes increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 3 | 0
Platelet count increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Transverse sinus thrombosis (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Elective surgery (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 0
Plastic surgery (Surgical and medical procedures) | 1 | 0
Skin cosmetic procedure (Surgical and medical procedures) | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Subgaleal haematoma (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim in Adults (N=291) | Romiplostim in Pediatric Population (N=20)
Anaemia (Blood and lymphatic system disorders) | 17 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 29 | 2
Abdominal discomfort (Gastrointestinal disorders) | 17 | 1
Abdominal pain (Gastrointestinal disorders) | 33 | 3
Abdominal pain upper (Gastrointestinal disorders) | 21 | 4
Constipation (Gastrointestinal disorders) | 26 | 1
Diarrhoea (Gastrointestinal disorders) | 72 | 2
Dyspepsia (Gastrointestinal disorders) | 19 | 0
Gingival bleeding (Gastrointestinal disorders) | 43 | 5
Mouth haemorrhage (Gastrointestinal disorders) | 21 | 4
Mouth ulceration (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 69 | 4
Toothache (Gastrointestinal disorders) | 17 | 1
Vomiting (Gastrointestinal disorders) | 46 | 7
Asthenia (General disorders) | 22 | 0
Chest pain (General disorders) | 16 | 1
Chills (General disorders) | 12 | 2
Fatigue (General disorders) | 93 | 7
Injection site haematoma (General disorders) | 15 | 0
Oedema peripheral (General disorders) | 41 | 0
Pain (General disorders) | 32 | 4
Pyrexia (General disorders) | 36 | 9
Seasonal allergy (Immune system disorders) | 16 | 1
Bronchitis (Infections and infestations) | 22 | 1
Ear infection (Infections and infestations) | 11 | 2
Gastroenteritis (Infections and infestations) | 13 | 2
Influenza (Infections and infestations) | 23 | 0
Nasopharyngitis (Infections and infestations) | 100 | 5
Sinusitis (Infections and infestations) | 38 | 1
Upper respiratory tract infection (Infections and infestations) | 76 | 10
Urinary tract infection (Infections and infestations) | 36 | 0
Viral infection (Infections and infestations) | 5 | 2
Viral upper respiratory tract infection (Infections and infestations) | 7 | 3
Animal bite (Injury, poisoning and procedural complications) | 3 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 88 | 8
Excoriation (Injury, poisoning and procedural complications) | 10 | 3
Fall (Injury, poisoning and procedural complications) | 19 | 0
Joint sprain (Injury, poisoning and procedural complications) | 11 | 2
Procedural pain (Injury, poisoning and procedural complications) | 17 | 2
Skin laceration (Injury, poisoning and procedural complications) | 18 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 16 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 29 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 55 | 2
Dizziness (Nervous system disorders) | 51 | 2
Headache (Nervous system disorders) | 109 | 9
Migraine (Nervous system disorders) | 15 | 1
Paraesthesia (Nervous system disorders) | 28 | 0
Anxiety (Psychiatric disorders) | 21 | 0
Depression (Psychiatric disorders) | 19 | 0
Insomnia (Psychiatric disorders) | 41 | 0
Dysuria (Renal and urinary disorders) | 15 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 70 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 73 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 30 | 6
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 20 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 50 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 5
Blood blister (Skin and subcutaneous tissue disorders) | 19 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 25 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 53 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 0
Rash (Skin and subcutaneous tissue disorders) | 44 | 5
Scab (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 18 | 1
Haematoma (Vascular disorders) | 37 | 1
Hypertension (Vascular disorders) | 17 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.